CLINICAL TRIAL: NCT02142153
Title: F901318 - A Phase I, Double-Blind, Placebo Controlled, Single Ascending Intravenous Dose, Safety, Tolerability and Pharmacokinetic Study in Healthy Male Subjects
Brief Title: F901318 Single Ascending Dose Study in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: F2G Biotech GmbH (Industry)
Collaborators: Simbec Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: F901318-01-01-14; 2014-000823-25 (EudraCT Number)
Record Dates: First submitted 2014-05-13; First posted 2014-05-20 (Estimated); Results first posted 2015-09-07 (Estimated); Last update posted 2015-09-07 (Estimated); Status verified 2015-06

CONDITIONS: Invasive Aspergillosis
Keywords: First in man; Antifungal; Intravenous infusion; Healthy volunteers
MeSH Terms: interventions — olorofim

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (10):
- F901318 0.25 mg/kg (Experimental): Single intravenous infusion over 4 hours
  Interventions: Drug: F901318
- 0.25 mg/kg placebo (Placebo Comparator): Single intravenous infusion over 4 hours
  Interventions: Drug: Placebo
- F901318 0.75 mg/kg (Experimental): Single intravenous infusion over 4 hours
  Interventions: Drug: F901318
- Placebo 0.75 mg/kg (Placebo Comparator): Single intravenous infusion over 4 hours
  Interventions: Drug: Placebo
- F901318 1.5 mg/kg (Experimental): Single intravenous infusion over 4 hours
  Interventions: Drug: F901318
- Placebo 1.5 mg/kg (Placebo Comparator): Single intravenous infusion over 4 hours
  Interventions: Drug: Placebo
- F901318 mg/kg (Experimental): Single intravenous infusion over 4 hours
  Interventions: Drug: F901318
- Placebo 3 mg/kg (Placebo Comparator): Single intravenous infusion over 4 hours
  Interventions: Drug: Placebo
- F901318 5 mg/kg (Experimental): Single intravenous infusion over 4 hours
  Interventions: Drug: F901318
- Placebo 5 mg/kg (Placebo Comparator): Single intravenous infusion over 4 hours
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: F901318 — Comparison of adverse events, clinically significant safety laboratory abnormalities and ECG abnormalities.
  Pharmacokinetic profile
  Arms: F901318 0.25 mg/kg; F901318 0.75 mg/kg; F901318 1.5 mg/kg; F901318 5 mg/kg; F901318 mg/kg
Drug: Placebo — Comparison of adverse events and clinically sign significant safety lab and ECG abnormalities
  Arms: 0.25 mg/kg placebo; Placebo 0.75 mg/kg; Placebo 1.5 mg/kg; Placebo 3 mg/kg; Placebo 5 mg/kg

SUMMARY:
F901318 is a potent new antifungal agent for the treatment of systemic fungal infections. This study will test it for the first time in man with the objective of assessing its safety, tolerability and pharmacokinetic profile.

DETAILED DESCRIPTION:
Double blind, placebo controlled, ascending single intravenous dose, sequential group study. Forty subjects will be studied in 5 cohorts (Groups A to E), each group consisting of 8 subjects. Each subject will be on study for approximately 6 weeks. Each subject will participate in one treatment cohort only, residing at the Clinical Research Unit (CRU) from Day -1 (the day before dosing) to Day 6 (120 hours post-dose). Each cohort will be dosed in a leading edge design in which two subjects will receive study drug (1 active and 1 placebo) on the first dosing day, and the last 6 will receive study drug (active or placebo) on the second dosing day.

All subjects will return for a post-study visit 8 to 10 days after the dose of study medication.

Cohorts will be dosed at 2 weekly intervals. There will be a review of safety and pharmacokinetic data prior to each dose escalation.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects will be males of any ethnic origin between 18 and 45 years of age and weighing 60-90 kg inclusive
2. Subjects must be in good health, as determined by a medical history, physical examination, 12-lead electrocardiogram (ECG) and clinical laboratory evaluations (congenital non haemolytic hyperbilirubinaemia is acceptable)
3. Subjects will have given their written informed consent to participate in the study and to abide by the study restrictions

Exclusion Criteria:

1. Male subjects who are not, or whose partners are not willing to use appropriate contraception (such as a condom) with established use of oral, injected or implanted hormonal contraceptive, intrauterine device or diaphragm with spermicide for three months after the last dose
2. Subjects who have received any prescribed systemic or topical medication within 14 days of dosing with study drug unless in the opinion of the Investigator and the Medical Monitor the medication will not interfere with the study procedures or compromise safety
3. Subjects who have used any non-prescribed systemic or topical medication (including herbal remedies) within 7 days of dosing with study drug (with the exception of vitamin/mineral supplements) unless in the opinion of the Investigator and the Medical Monitor the medication will not interfere with the study procedures or compromise safety
4. Subjects who have received any medications, including St John's Wort, known to chronically alter drug absorption or elimination processes within 30 days of dosing with study drug unless in the opinion of the Investigator and the Medical Monitor the medication will not interfere with the study procedures or compromise safety
5. Subjects who are still participating in a clinical study (e.g. attending follow-up visits) or who have participated in a clinical study involving administration of an investigational drug (new chemical or biological entity) in the past 3 months

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2014-08; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Salvatore Febbraro, MD, Principal Investigator — Simbec Research
Locations (1):
- Simbec Research, Merthyr Tydfil, Mid Glamorgan, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- F901318 0.25 mg/kg; F901318 0.75 mg/kg; F901318 1.5 mg/kg; F901318 3 mg/kg; F901318 4 mg/kg: Single intravenous infusion over 4 hours
  F901318: Comparison of adverse events, clinically significant safety laboratory abnormalities and ECG abnormalities.
  Pharmacokinetic profile
- Placebo 4 mg/kg: Single intravenous infusion over 4 hours
  Placebo: Comparison of adverse events and clinically sign significant safety lab and ECG abnormalities
Period: Overall Study
Arm/Group | F901318 0.25 mg/kg | 0.25 mg/kg Placebo | F901318 0.75 mg/kg | Placebo 0.75 mg/kg | F901318 1.5 mg/kg | Placebo 1.5 mg/kg | F901318 3 mg/kg | Placebo 3 mg/kg | F901318 4 mg/kg | Placebo 4 mg/kg
Started | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2
Completed | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Healthy volunteers
Groups:
- Total: Total of all reporting groups
Arm/Group | F901318 0.25 mg/kg | 0.25 mg/kg Placebo | F901318 0.75 mg/kg | Placebo 0.75 mg/kg | F901318 1.5 mg/kg | Placebo 1.5 mg/kg | F901318 3 mg/kg | Placebo 3 mg/kg | F901318 4 mg/kg | Placebo 4 mg/kg | Total
Number analyzed (Participants) | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 40
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 40
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 40

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Adverse Events
Description: Adverse events will be collected from the time of screening until the final study visit
Time Frame: Single dose
Population: Full analytical set
Measure: Number; unit: participants
Arm/Group | F901318 0.25 mg/kg | 0.25 mg/kg Placebo | F901318 0.75 mg/kg | Placebo 0.75 mg/kg | F901318 1.5 mg/kg | Placebo 1.5 mg/kg | F901318 3 mg/kg | Placebo 3 mg/kg | F901318 4 mg/kg | Placebo 4 mg/kg
Number analyzed (Participants) | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2
participants | 1 | 1 | 1 | 1 | 1 | 0 | 1 | 0 | 1 | 0

2. Secondary Outcome: Number of Subjects With Significant Clinical Safety Labs and ECG Abnormalities
Description: Number of subjects with significant Clinical safety labs and ECG abnormalities as judged by the investigator from screening until final study visit
Time Frame: Single dose
Measure: Number; unit: participants
Groups:
- F901318 0.25 mg/kg; F901318 0.75 mg/kg; F901318 1.5 mg/kg; F901318 3 mg/kg; F901318 4 mg/kg: Single intravenous infusion over 4 hours
  F901318: Comparison of clinically significant safety laboratory abnormalities and ECG abnormalities.
  No clinically significant findings
- 0.25 mg/kg Placebo: Single intravenous infusion over 4 hours
  Placebo: Comparison of clinically significant safety lab and ECG abnormalities No clinically significant findings
- Placebo 0.75 mg/kg; Placebo 1.5 mg/kg; Placebo 3 mg/kg; Placebo 4 mg/kg: Single intravenous infusion over 4 hours
  Placebo: Comparison of clinically sign significant safety lab and ECG abnormalities No clinically significant findings
Arm/Group | F901318 0.25 mg/kg | 0.25 mg/kg Placebo | F901318 0.75 mg/kg | Placebo 0.75 mg/kg | F901318 1.5 mg/kg | Placebo 1.5 mg/kg | F901318 3 mg/kg | Placebo 3 mg/kg | F901318 4 mg/kg | Placebo 4 mg/kg
Number analyzed (Participants) | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2
participants | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2

3. Other Pre Specified Outcome: Pharmacokinetics
Description: Blood samples (6 mL) for analysis of F901318 plasma concentration will be drawn pre-dose and at 1h, 2h, 3h and 4h and then 4.25, 4.5, 5.0, 5.5, 6, 7, 8, 10, 12, 24, 36, 48, 72, 96 and 120 hours following the start of the infusion. (20 samples).
Time Frame: Single dose
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 120 hours
Arm/Group | F901318 0.25 mg/kg | 0.25 mg/kg Placebo | F901318 0.75 mg/kg | Placebo 0.75 mg/kg | F901318 1.5 mg/kg | Placebo 1.5 mg/kg | F901318 3 mg/kg | Placebo 3 mg/kg | F901318 4 mg/kg | Placebo 4 mg/kg
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/2 | 0/6 | 0/2 | 0/6 | 0/2 | 0/6 | 0/2 | 0/6 | 0/2
Other Adverse Events (participants affected / at risk) | 1/6 | 1/2 | 1/6 | 1/2 | 1/6 | 0/2 | 1/6 | 0/2 | 1/6 | 0/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | F901318 0.25 mg/kg (N=6) | 0.25 mg/kg Placebo (N=2) | F901318 0.75 mg/kg (N=6) | Placebo 0.75 mg/kg (N=2) | F901318 1.5 mg/kg (N=6) | Placebo 1.5 mg/kg (N=2) | F901318 3 mg/kg (N=6) | Placebo 3 mg/kg (N=2) | F901318 4 mg/kg (N=6) | Placebo 4 mg/kg (N=2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Epistaxis
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Pareasthesia
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Pain in extremity
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Headache
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Eczema

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No